CLINICAL TRIAL: NCT06324253
Title: Comparison of Thoracic Epidural Analgesia With Ultrasound-Guided Bilateral Erector Spinae Plane Block in Radical Cystectomy Surgery: A Randomised Trial
Brief Title: Thoracic Epidural Analgesia With Bilateral Erector Spinae Plane Block in Radical Cystectomy Surgery
Acronym: TEAvsESB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Collaborators: Amal Ismael Abdelrahman Hassan (Unknown); Ibrahim Mowafy Gomaa Atawia (Unknown)
Responsible Party: Principal Investigator, Amal Gouda Elsayed Safan, lecturer of anaethesia, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1/24 UROL2
Record Dates: First submitted 2024-01-26; First posted 2024-03-21 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Tea

STUDY DESIGN:
Intervention Model Description: Group A: will receive bilateral Erector Spinae Block after induction of anesthesia.
  Group B: will receive Thoracic Epidural Block before induction of anesthesia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Block (Active Comparator): after induction of anesthesia bilateral US ESP block will be performed in the left lateral decubitus position under strict aseptic precautions. linear ultrasound transducer will be placed in a sterile cover, and positioned on the midline to identify the T10 spinous process. From this position, the ultrasound transducer will be moved 2-3 cm laterally to visualise the hyperechoic line of the T10 transverse process with its associated acoustic shadow inferiorly, and the overlying erector spinae muscle superiorly. Using in-plane approach a needle will be inserted in caudal-cephalad direction, until the tip is contact with the T10 transverse process and will be in the interfacial plane deep to the erector spinae muscle group and A dose of 30 ml 0.125% Bupivacaine will be injected bilateral in this plane . All patients will receive 1g intravenous paracetamol and 4 grams ondansetron 8mg dexamethasone
  Interventions: Procedure: bilateral Erector spine block,A dose of 30 ml 0.125% Bupivacaine will be injected.
- Thoracic Epidural Block (Active Comparator): before induction of anesthesia under strict aseptic precautions, 18Gauge Tuohy's needle with Huber's tip will be inserted via median approach after local infiltration with 5 ml of 2% lignocaine at the level of T9-T10 or T10-T11 intervertebral space in the sitting position. After identifying epidural space using loss of resistance technique, 5 ml of saline will be administered after negative aspiration for blood or cerebrospinal fluid and 20Gauge epidural catheter will be threaded 5 cm cranially.
  the patients in group B will be administered with a bolus dose of 10 ml of 0.125% bupivacaine through epidural catheter followed by continuous infusion of 0.125% bupivacaine at the rate of 0.1 ml/kg/hour All patients will receive 1g intravenous paracetamol and 4 grams ondansetron 8mg dexamethasone
  Interventions: Procedure: Thoracic epidural analgesia

INTERVENTIONS:
Procedure: bilateral Erector spine block,A dose of 30 ml 0.125% Bupivacaine will be injected. — will receive bilateral Erector Spinae Block after induction of anesthesia
  Other Names: ESB
  Arms: Erector Spinae Block
Procedure: Thoracic epidural analgesia — will receive Thoracic Epidural Block before induction of anesthesia .a bolus dose of 10 ml of 0.125% bupivacaine through epidural catheter followed by continuous infusion of 0.125% bupivacaine at the rate of 0.1 ml/kg/hour
  Other Names: TEA
  Arms: Thoracic Epidural Block

SUMMARY:
The aim of this study is to compare between Thoracic Epidural Analgesia (TEA) with ultrasound-guided bilateral erector spinae plane (ESP) block in radical cystectomy surgery for analgesic efficacy and hemodynamic effects

DETAILED DESCRIPTION:
The patients will be randomly allocated into two equal groups using a computer program.

Group A: will receive bilateral Erector Spinae Block after induction of anesthesia.

Group B: will receive Thoracic Epidural Block before induction of anesthesia.

The methods:

Preoperative evaluation of each patient will include full history taking, revision of all laboratory investigations and full clinical examination.

On arrival to the operation room, a standard monitoring will be connected to the patient

In group A, after induction of anesthesia bilateral Ultrasound ESP block will be performed in the left lateral decubitus position under strict aseptic precautions. linear ultrasound transducer will be placed in a sterile cover, and positioned on the midline to identify the T10 spinous process. From this position, the ultrasound transducer will be moved 2-3 cm laterally to visualise the hyperechoic line of the T10 transverse process with its associated acoustic shadow inferiorly, and the overlying erector spinae muscle superiorly. transverse using in-plane approach a needle will be inserted in caudal-cephalad direction, until the tip is contact with the T10 transverse process and will be in the interfacial plane deep to the erector spinae muscle group. A dose of 30 ml 0.125% Bupivacaine will be injected.

In group B, before induction of anesthesia under strict aseptic precautions, 18Gauge Tuohy's needle with Huber's tip will be inserted via median approach after local infiltration with 5 ml of 2% lignocaine at the level of T9-T10 or T10-T11 intervertebral space in the sitting position. After identifying epidural space using loss of resistance technique, 5 ml of saline will be administered after negative aspiration for blood or cerebrospinal fluid and 20Gauge epidural catheter will be threaded 5 cm cranially.then will be administered a bolus dose of 10 ml of 0.125% bupivacaine through epidural catheter followed by continuous infusion of 0.125% bupivacaine at the rate of 0.1 ml/kg/hour . Patients in either group with inadequate analgesia will be excluded from the study.

General anesthesia induction will be achieved using fentanyl 1µg/kg (IV), propofol 2mg/kg (IV), and0.5mg/kg of IV Atracurium. General anesthesia will be maintained with mechanical ventilation with isoflurane (MAC 0.8: 1.2) with O2 \ Air mixture.

During anesthesia maintenance Intraoperatively, if BP or heart rate (HR) increase more than 20% from baseline, intravenous morphine will be given to stabilize the patients' haemodynamics.

All patients will receive 1g intravenous paracetamol and 4 grams ondansetron 8mg dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

- Eligible patients will be older than 40-70 years old with american society of ASA physical anesthesiologist status I, II and III scheduled for elective radical cystectomy surgeries

Exclusion Criteria:

* Patients who have allergy to any of the study drugs.
* Patients who are on opioids.
* Known abuse of alcohol or medication.
* Local infection at the site of injection or systemic infection.
* Pregnancy
* Patients with coagulation disorders or on anticoagulation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Time for first rescue analgesia | 24 hours
  the time of request of the patient of analgesia wil be recorded

SECONDARY OUTCOMES:
Visual analogue scale score at 1st,2nd,4th,6th,8th,12th and 24 h (where 0 is interpreted as no pain, 1-4 mild pain, 5-6 moderate pain, 7-10 severe pain) | 24 hours
  the record of patient expression to pain wil be recorded
the number of rescue analgesics within 24hrs after surgery | 24 hours
  total opioid consumption

OTHER OUTCOMES:
The heart rate, mean arterial blood pressure | pulse per minute--mmhge
  the HR and MBP will be recorded perioperative
Complications like bradycardia or hypotension, intraoperative and postoperative dysrhythmia, nausea and vomiting | 24 hours
  possible complications to the blocks wil be recorded

CONTACTS AND LOCATIONS:
Overall Officials: AMAL G SAFAN, MD, Principal Investigator — Menoufia University
Locations (1):
- Menoufia university, Cairo, Shibin Elkom, Egypt